CLINICAL TRIAL: NCT01918306
Title: A Phase Ib/II Trial of GDC-0941 (a PI3K Inhibitor) in Combination With Cisplatin in Patients With Androgen Receptor Negative Triple Negative Metastatic Breast Cancer
Brief Title: GDC-0941 and Cisplatin in Treating Patients With Androgen Receptor-Negative Triple Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: company stopped production of study drug due to excessive toxicities, lack of efficacy
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Vandana Abramson, Assistant Professor of Medicine; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 1287; NCI-2013-01319 (Other: NCI)
Record Dates: First submitted 2013-07-25; First posted 2013-08-07 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Estrogen Receptor Negative Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Triple Negative Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer; Triple-negative Breast Cancer
Keywords: Triple Negative Breast Cancer; Estrogen receptor negative breast cancer; Metastatic breast cancer; Stage IV breast cancer; HER2 negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Cisplatin; 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1PHIbA Arm A - cisplatin + GDC - 0941 (Experimental): Determine the safety and tolerability of GDC-0941 given in combination with cisplatin in patients with AR- TN MBC. Determination of the maximally tolerated dose (MTD) of GDC-0941.
  Cohort 1, 3 of 3 patients received:
  Cisplatin 25 mg/m2 IV D1, 8, 15 GDC-0941 260 mg PO, days 2-6, 9-13, 16-20, 23-27, 28 day cycle GDC-0941 dose to start at Max dose of 260mg.
  If no patient in the first cohort of 3 experiences a DLT, an additional cohort of 3 patients will be treated at the same dose level.
  1. If 1 patient experiences a DLT in the first cohort, an additional cohort of 3 patients will be treated at the same dose level.
  2. If ≤1 patient has a DLT in 6 treated at this same dose, this will be considered a tolerable dose to move to phase II
  If patients experience a DLT considered related to GDC-0941, the patient may remain on GDC-0941 and/or Cisplatin after resolution of the DLT. All such cases will be considered a DLT for the purposes of defining the MTD.
  Interventions: Drug: cisplatin; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI; Drug: GDC -0941
- 1PHIbB - Arm B - Cisplatin + GDC 0941 dose level -1 (Experimental): If 2 or more patients in 3 or 6 patients treated at a given dose experience DLT, the dose will be de-escalated to the next lower dose level. Once the lowest dose level is reached, if a DLT occurs, the regimen will be considered too toxic and the corresponding cohort within the study will be discontinued.
  Determination of the maximally tolerated dose (MTD) of GDC-0941.
  Interventions: Drug: cisplatin; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI; Drug: GDC -0941
- 2PHII1 Arm 1 - Cisplatin (Active Comparator): Evaluate the efficacy, as measured by the overall response rate (ORR), of Cisplatin +GDC-0941 versus Cisplatin alone in patients with AR- TN MBC.
  Patients will be randomized in a 1:1 fashion to arm 1: cisplatin, or arm 2: cisplatin + GDC-0941.
  Arm 1 Cisplatin Only Patient received:
  Cisplatin given intravenously (IV) over 1 hour for three consecutive weeks, then off one week (days 1, 8, and 15 of a 28 day cycle).
  Interventions: Drug: cisplatin; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI
- 2PHII2 - Arm 2 - Cisplatin + GDC - 0941 (Experimental): Evaluate the efficacy, as measured by the overall response rate (ORR), of Cisplatin +GDC-0941 versus Cisplatin alone in patients with AR- TN MBC. Patients are randomized in a 1:1 fashion to arm 1: cisplatin, or arm 2: cisplatin + GDC-0941.
  Arm 2 Cisplatin + GDC-0941 Patients received:
  Cisplatin given intravenously (IV) over 1 hour for three consecutive weeks, then off one week (days 1, 8, and 15 of a 28 day cycle).
  GDC-0941 260 mg PO, administered orally on days 2-6, 9-13, 16-20, 23-27 of a 28 day cycle.
  Interventions: Drug: cisplatin; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI; Drug: GDC -0941
- 2PHIICO (Experimental): Arm 2: Crossover post-progression
  Patients who are randomized to Cisplatin alone (Arm 1) can crossover to receive Cisplatin + GDC-0941 upon disease progression.
  Patient received:
  Cisplatin given intravenously (IV) over 1 hour for three consecutive weeks, then off one week (days 1, 8, and 15 of a 28 day cycle).
  GDC-0941 260 mg PO, administered orally on days 2-6, 9-13, 16-20, 23-27 of a 28 day cycle.
  Interventions: Drug: cisplatin; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI; Drug: GDC -0941

INTERVENTIONS:
Drug: cisplatin — In Arm I patients receive cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may crossover to Arm II upon disease progression.
  In Arm II patients receive cisplatin as in Arm I and PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  --------------------------------------------------------------------------------
  Other Names: Platinol
Other: laboratory biomarker analysis — correlative studies
Other: pharmacological study — correlative studies
Procedure: dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI — correlative studies
Drug: GDC -0941 — Patients receive cisplatin as in Arm I and PI3K inhibitor GDC-0941 PO QD on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Arms: 1PHIbA Arm A - cisplatin + GDC - 0941; 1PHIbB - Arm B - Cisplatin + GDC 0941 dose level -1; 2PHII2 - Arm 2 - Cisplatin + GDC - 0941; 2PHIICO

SUMMARY:
This phase I/II trial study evaluates the tolerability and best tolerated dose of the PI3K inhibitor GDC-0941 when given with the chemotherapy cisplatin. This study will also examine how well the combination of GDC-0941 and cisplatin work in treating patients with androgen receptor negative triple negative metastatic breast cancer. Patients will be randomized to receive cisplatin alone or cisplatin with GDC-0941 in the phase II portion. Those receiving cisplatin alone can receive GDC-0941 upon progression of their disease. Cisplatin is a chemotherapy which has been shown to be effective in treating triple negative breast cancer. Preclinical studies show that adding a PI3K inhibitor such as GDC-0941 to cisplatin may be a more effective treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of GDC-0941 when given in combination with cisplatin in patients with androgen receptor-negative (AR-) triple negative (TN) metastatic breast cancer (MBC): assessment of dose limiting toxicities (DLTs) during the first 4 weeks of treatment (cycle 1); determination of the maximally tolerated dose (MTD) and recommended phase II dose of GDC-0941 given in combination with cisplatin. (Phase IB)

II. To evaluate the efficacy, as measured by the overall response rate (ORR), of cisplatin + GDC-0941 versus cisplatin alone in patients with AR- TN MBC. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the clinical benefit rate (CBR) of cisplatin + GDC-0941 in patients with AR- TN MBC.

II. To determine the time to disease progression (TTP) of cisplatin + GDC-0941 versus cisplatin alone in patients with AR- TN MBC.

TERTIARY OBJECTIVES:

I. To characterize pharmacokinetics of GDC-0941 when administered in combination with cisplatin.

II. To explore predictors of response and mechanisms of resistance based on exploratory analysis of tumor tissue obtained through biopsies.

III. To assess the prognostic effects of phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutations and phosphatase and tensin homolog (PTEN) loss on TTP and CBR.

OUTLINE: This is a phase I, dose-deescalation study of PI3K inhibitor GDC-0941 followed by a randomized phase II study.

PHASE I: Patients receive cisplatin intravenously (IV) over 1 hour on days 1, 8, and 15 and PI3K inhibitor GDC-0941 orally (PO) once daily (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may crossover to Arm II upon disease progression.

ARM II: Patients receive cisplatin as in Arm I and PI3K inhibitor GDC-0941 PO QD on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide informed written consent.
* Patients must be <18 years of age.
* ECOG performance status 0-1.
* Clinical stage IV invasive mammary carcinoma, ER negative (defined as expression of ER in < 5% cells), PR negative (defined as expression of PR in < 5% cells), HER2 negative [acceptable FDA approved methods of HER2 analysis include IHC (0, 1+), fluorescence in situ hybridization (FISH) with HER2/CEN-17 ratio <2, and/or chromogenic in situ hybridization (CISH)] with HER2/CEN-17 ratio <2, as previously documented by histological analysis.
* Androgen receptor negativity, defined as < 10% of tumor cell nuclei with immunoreactivity for AR in a CLIA certified laboratory. See section 5.1.
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension by RECIST criteria 1.1, with radiologic scans within 21 days of day 1, cycle 1.
* Up to one prior chemotherapy regimens for metastatic disease.
* No prior treatment with cisplatin in the metastatic setting.
* Biopsy of a metastatic lesion in patients with reasonably accessible metastatic lesions (chest wall, skin, subcutaneous tissue, lymph nodes, skin, breast, bones, lung, and liver metastases). If a reasonably accessible site is available for biopsy, the patient must agree to biopsy.
* Life expectancy ≥ 6 months in the opinion of the investigator
* Patients must have adequate hematologic, hepatic, and renal function. All tests must be obtained less than 21 days from day 1 of study treatment. This includes:

  * ANC >/=1500/mm3
  * Platelet count >/=100,000/mm3
  * Hemoglobin ≥ 9 g/dL
  * Creatinine </=1.5X upper limits of normal (ULN)
  * INR ≤ 2
  * Total serum bilirubin ≤ 1.5 x ULN (in patients with known Gilbert Syndrome, a total bilirubin ≤ 3.0 x ULN, with direct bilirubin ≤ 1.5 x ULN)
  * AST and ALT ≤ 3 x ULN (or ≤ 5.0 x ULN if hepatic metastases are present)
  * For patients without known Type II diabetes, the following is required at screening:

    o -Fasting blood glucose </= 135 mg/dL (7.49 mmol/L) and glycosylated hemoglobin (HbA1c) <7.0 % or International Federation of Clinical Chemistry (IFCC) < 53 mmol/mol
  * For patients with Type II diabetes receiving only oral anti-hyperglycemic therapy (patients receiving insulin are not eligible), the following are required at screening:

    * -HbA1c < 8.5 % or IFCC < 69.4 mmol/mol
    * -Stable regimen of oral anti-hyperglycemic therapy without insulin usage for at least 3 weeks prior to first study treatment
    * -Fasting blood glucose levels </= 160 mg/dL (8.88 mmol/L) and no hypoglycemia (BS <60) during home monitoring for at least 1 week prior to study entry
* Patients must be able to swallow and retain oral medication.
* For patients who are not postmenopausal or surgically sterile (absence of ovaries and/or uterus), agreement to remain abstinent or to use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year (e.g., hormonal implants, combined oral contraceptives, vasectomy/vasectomized partner, tubal ligation), during the treatment period and for at least 30 days after the last dose of GDC-0941 or 6 months after the last dose of cisplatin, whichever is longer; postmenopausal is defined as:
* Age >/= 60 years
* Age </= 60 years and amenorrheic for 12 months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression; and follicle stimulating hormone and estradiol in the postmenopausal range
* Patients may have received radiation therapy to painful bone metastases or areas of impending bone fracture as long as radiation therapy is completed ≥ 2 weeks prior to day 1 of cycle 1 of treatment. Patients who have received prior radiotherapy must have recovered from toxicity (≤ grade 1) induced by this treatment. Baseline radiologic scans must be obtained after completion of radiation.
* Patients must complete all screening assessments as outlined in the protocol.

Exclusion Criteria:

* Any kind of malabsorption syndrome significantly affecting gastrointestinal function.
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, biologic therapy) other than the ones specified in the protocol. Patients must have discontinued the above cancer therapies for 1 week prior to the first dose of study medication, as well as recovered from toxicity (to ≤ than grade 1, except for alopecia) induced by previous treatments. Any investigational drugs should be discontinued 2 weeks prior to the first dose of study medication and radiotherapy must have been completed ≥ 2 weeks prior to initiation of study drug (Cycle 1, Day 1).
* Prior use of PI3K, or Akt inhibitors in the neoadjuvant, adjuvant, and metastatic setting for the treatment of cancer. These include, but are not limited to: GDC-0941, GDC-0980, GDC-0032, BEZ235, BKM120, LY294002, PIK-75, TGX-221, XL147, XL765, SF1126, PX-866, D-87503, D-106669, GSK615, CAL101. Patients who have received PI3K/Akt inhibitors previously for <4 weeks will be eligible.
* Pregnant or lactating women.
* Insulin-dependent diabetes. Patients with Type II diabetes must meet criteria outlined in Inclusion Criteria.
* Uncontrolled intercurrent illness including, but not limited to:

  * -Ongoing or active infection requiring parenteral antibiotics
  * -Impairment of lung function (COPD > grade 2, lung conditions requiring oxygen therapy) or current dyspnea at rest
  * -Symptomatic congestive heart failure (class III or IV of the New York Heart Association classification for heart disease)
  * -Known Left Ventricular Ejection Fraction (LVEF) < 50%.
  * -Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
  * -Uncontrolled hypertension (systolic blood pressure >160 mm Hg or diastolic blood pressure > 100 mm Hg, found on two consecutive measurements separated by a 1 or 2 week period despite adequate medical support)
  * -Clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment [National Cancer Institute -Common Terminology Criteria for Adverse Events, Version 4.0, grade 3]
  * -QTcF ≥ 480 msec on screening EKG
  * -Known history of QT/QTc prolongation or Torsades de Pointes (TdP)
  * -ST depression or elevation of ≥ 1.5 mm in 2 or more leads
  * -Diarrhea of any cause ≥ CTCAE grade 2
  * -Active autoimmune disease that is not controlled by nonsteroidal or steroidal (<10 mg of prednisone per day) anti inflammatory drugs or active inflammatory disease, including small or large intestine inflammation such as active Crohn's disease or ulcerative colitis, which requires immunosuppressive therapy
  * -Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements including maintenance of a compliance/pill diary
  * -Symptomatic brain metastases (patients with a history of brain metastases must be clinically stable for at least 2 weeks from completion of radiation treatment, on a dose of steroids equivalent to <10 mg prednisone daily for at least one week, and on a stable dose of therapeutic anticonvulsants)
  * -Known history of chronic liver disease, including cirrhosis, current alcohol abuse, or infection with hepatitis B virus or hepatitis C virus (active or carrier), or renal failure
  * -Known history of chronic pancreatitis
  * -Conditions that affect lymphocyte counts, such as HIV infection or immunosuppressive therapy
* Use of prohibited drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vandana G. Abramson, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina, Charlotte, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor Breast Center, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial opened to accrual on 9/23/2013 and closed to accrual on 3/9/2016.
Groups:
- 1PHIbA - Arm A - Cisplatin + GDC -0941 Dose Level 1 Cohort 1&2: Patients receive cisplatin and PI3K inhibitor GDC-0941. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients receive cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor: GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- 1PHIbB - Arm B - Cisplatin + GDC -0941 Dose Level -1: If 2 or more patients in 3 or 6 patients (cohort 1 and 2) treated at a given dose 260 mg experience DLT, the dose will be de-escalated to the next lower dose level.
- 2PHII1 - Arm 1 - Cisplatin Only: Patients receive cisplatin in Arm I. Patients may crossover to Arm II upon disease progression.
  cisplatin: In Arm I patients receive cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may crossover to Arm II upon disease progression.
  --------------------------------------------------------------------------------
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
- 2PHII2 - Arm 2 - Cisplatin and GDC-0941: Patients receive Cisplatin and PI3K inhibitor GDC-0941. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients received cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  patients receive PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
Period: Overall Study
Arm/Group | 1PHIbA - Arm A - Cisplatin + GDC -0941 Dose Level 1 Cohort 1&2 | 1PHIbB - Arm B - Cisplatin + GDC -0941 Dose Level -1 | 2PHII1 - Arm 1 - Cisplatin Only | 2PHII2 - Arm 2 - Cisplatin and GDC-0941
Started (11 total patients. 2 pts received Cisplatin alone. 9 pts started Cisplatin and GDC-0941.) | 6 | 0 (No patients enrolled) | 2 (1 participant Crossed-over to ARM 2) | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 2 | 3
Not completed — progresive disease | 4 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — neutropenia | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — progress disease, crossover | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant that is listed in Cisplatin and GDC-0941 arm is a Crossover patient from the Cisplatin only arm.
Groups:
- Cisplatin: Patients receive cisplatin in Arm I. Patients may crossover to Arm II upon disease progression.
  cisplatin: In Arm I patients receive cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may crossover to Arm II upon disease progression.
  In Arm II patients receive cisplatin as in Arm I and PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  --------------------------------------------------------------------------------
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
- Cisplatin and GDC-0941: Patients receive cisplatin as in Arm I and PI3K inhibitor GDC-0941. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: In Arm I patients receive cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may crossover to Arm II upon disease progression.
  In Arm II patients receive cisplatin as in Arm I and PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  --------------------------------------------------------------------------------
  GDC -0941: Patients receive cisplatin as in Arm I and PI3K inhibitor GDC-0941 PO QD on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
- Total: Total of all reporting groups
Arm/Group | Cisplatin | Cisplatin and GDC-0941 | Total
Number analyzed (Participants) | 2 | 9 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 9 | 10
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (15.556) | 51.3 (10.1000) | 53.08 (11.081)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 9 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose(MTD) of GDC-0941 and Recommended Phase II Dose of GDC-0941 Given in Combination With Cisplatin. - (Phase Ib)
Description: GDC-0941 dose will start at 260 mg (maximum dose). De-escalation of the intensity of the dose (if necessary) will proceed among cohorts of 3 patients according to a standard 3+3 algorithm beginning at the highest dose level of GDC-0941 260mg.
  MTD is defined as the highest dose at which a DLT is experienced >= 1 out of 6 patients.
  A cohort of 3 patients was initially enrolled in the GDC-0941 arm at dose 260mg PO days 2-6, 9-13, 16-20, 23-27 of 28 day cycle
  1. If no patient in the first cohort of 3 experiences a DLT, an additional cohort of 3 patients will be treated at the same dose level.
  2. If 1 patient experiences a DLT in the first cohort, an additional cohort of 3 patients will be treated at the same dose level.
  3. If ≤1 patient has a DLT in 6 treated at this same dose, this will be considered a tolerable dose to move to phase II.
  4. If 2 or more patients in 3 or 6 patients treated at a given dose experience DLT, the dose will be de-escalated to the next lower dose level.
Time Frame: 4 weeks
Population: A cohort of 3 was enrolled at dose 260mg. No DLT was found. Then a second cohort of 260mg was enrolled. One of them experienced DLT.
Measure: Number; unit: mg
Groups:
- 1PHIbA -Cisplatin and GDC-0941: Patients receive cisplatin and PI3K inhibitor GDC-0941. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients receive cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor: GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | 1PHIbA -Cisplatin and GDC-0941
Number analyzed (Participants) | 6
mg | 260

2. Primary Outcome: Percentage of Patients Achieving Overall Response - (Phase II)
Description: The primary efficacy endpoint is overall response rate (ORR) of cisplatin + GDC-0941 versus cisplatin alone in patients with AR- TN MBC. ORR is defined as the percentage of subjects achieving complete response (CR) plus partial response (PR) as their best response by RECIST version 1.1 for targeted lesions and assessed by CT, MRI scan.
  Objective responses, was estimated by the overall tumor burden at baseline (targeted lesions) in which subsequent measurements were performed every 8 weeks using the Solid Tumor Response Criteria (RECIST) v1.1 were compared. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: at 8 weeks
Population: Phase 1-Initial and Max tolerated dose of GCD-0941 was the same, no dose de-escalation occurred. Phase 2, 1 of the 2 patients from the Cisplatin only arm did crossover to the Crossover Cisplatin and GDC-0941 arm. 3 patients randomized to Cisplatin + GDC -0941 arm, and 1 crossover patient, for a total of 4 patients who received Cisplatin+GDC-0941.
Measure: Count of Participants; unit: Participants
Groups:
- 2PHII1 Arm 1 Cisplatin: Patients receive cisplatin in Arm I. Patients may crossover to Arm II upon disease progression.
  cisplatin:patients received cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may crossover to Arm II upon disease progression.
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
- 2PHII2 Arm 2 - Cisplatin and GDC-0941: Patients receive Cisplatin and PI3K inhibitor GDC-0941. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients received cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  patients receive PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
- 2PHIICO - Crossover to Arm 2 - Cisplatin and GDC-0941: Crossover patient received Cisplatin and PI3K inhibitor GDC-0941 after found to have disease progression in Cisplatin only arm. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients received cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  patients receive PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
Arm/Group | 2PHII1 Arm 1 Cisplatin | 2PHII2 Arm 2 - Cisplatin and GDC-0941 | 2PHIICO - Crossover to Arm 2 - Cisplatin and GDC-0941
Number analyzed (Participants) | 2 | 3 | 1
Participants | 0 | 1 | 0

3. Secondary Outcome: Number of Patients With Dose-limiting Toxicities Per NCI Common Terminology for Adverse Events (CTCAE) - (Phase Ib)
Description: Number of patients with Grade 3 and 4 toxicities per NCI Common Terminology for Adverse Events (CTCAE) version 4.0 requirements.
Time Frame: During the first 4 weeks
Population: Less than 2 patients in cohort 1 and 2 experienced DLT, therefore no patients enrolled in arm 1PHIbB.
Measure: Number; unit: participants
Groups:
- 1PHIbA - Cisplatin and GDC-0941 Cohort 1: Starting dose of GDC - 0941 260mg. De-escalation of the intensity of the dose (if necessary) will proceed among cohorts of 3 patients according to a standard 3+3 algorithm beginning at the highest dose level. (Highest dose = 260mg)
  In cohort 1 patients received Cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also received PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- 1 PHIbA - Arm 1 - Cisplatin and GDC-0941Cohort 2: Starting dose of GDC - 0941 260mg, no DLT's experienced in cohort 1. Therefore no de-escalation of the intensity of the dose was necessary. An additional cohort of 3 patients will be treated at the same dose level beginning at the highest dose level. (Highest dose = 260mg)
  In cohort 2, patients received Cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also received PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  ≤1 patient has a DLT in 6 treated at this same dose, this will be considered a tolerable dose to move to phase II.
- 1PHIbB - Arm B - Cistplatin + GDC -0941 Dose Level -1: If 2 or more patients in 3 or 6 patients (cohort 1 and 2) treated at a given dose 260 mg experience DLT, the dose will be de-escalated to the next lower dose level.
Arm/Group | 1PHIbA - Cisplatin and GDC-0941 Cohort 1 | 1 PHIbA - Arm 1 - Cisplatin and GDC-0941Cohort 2 | 1PHIbB - Arm B - Cistplatin + GDC -0941 Dose Level -1
Number analyzed (Participants) | 3 | 3 | 0
participants | 0 | 1 |

4. Secondary Outcome: Clinical Benefit Rate - (Phase II)
Description: Clinical Benefit Rate (CBR) is defined as complete response (CR) plus partial response (PR) plus stable disease (SD) for 6 months.
  Clinical Benefit Rate (CBR) is calculated with the corresponding 95% confidence intervals at the dose recommended for phase II.
  Response and progression will be evaluated using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 performed at baseline and every 8 weeks will be compared.
Time Frame: at 32 weeks
Population: Study closed early and response and progression were not evaluated at 32 weeks.
Groups:
- 2 PHII1 - ARM 1 Cisplatin: Patients receive Cisplatin in Arm I. Patients may crossover to Arm II upon disease progression.
  Cisplatin: patients received Cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may crossover to Arm II upon disease progression.
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
- 2PHIICO - Crossover to 2 - Cisplatin + GDC-0941: Crossover patient received Cisplatin and PI3K inhibitor GDC-0941 after found to have disease progression in Cisplatin only arm. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients received cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  patients receive PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
Arm/Group | 2 PHII1 - ARM 1 Cisplatin | 2PHII2 - ARM 2 - Cisplatin and GDC-0941 | 2PHIICO - Crossover to 2 - Cisplatin + GDC-0941
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

5. Secondary Outcome: Time to Progression - (Phase II)
Description: Time to Progression (TTP) is calculated with the corresponding 95% confidence interval at the dose recommended for phase II. TTP is defined as the time from randomization until objective tumor progression, this does not include deaths unrelated to disease progression.
Time Frame: From time of randomization to disease progression, up to 104 weeks
Measure: Median (Full Range); unit: days to progression
Groups:
- 2PHII1 - Arm 1 - Cisplatin: Patients receive Cisplatin in Arm I. Patients may crossover to Arm II upon disease progression.
  Cisplatin: patients received Cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may crossover to Arm II upon disease progression.
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
- 2PHIICO - Crossover to Arm 2 - Cistplatin + GDC - 0941: Crossover patient received Cisplatin and PI3K inhibitor GDC-0941 after found to have disease progression in Cisplatin only arm. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients received cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  patients receive PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
Arm/Group | 2PHII1 - Arm 1 - Cisplatin | 2PHII2 - Arm 2 - Cisplatin and GDC-0941 | 2PHIICO - Crossover to Arm 2 - Cistplatin + GDC - 0941
Number analyzed (Participants) | 2 | 3 | 1
days to progression | 24.5 [9 to 40] | NA [56 to 56] — 1 patient progressed at 56 days, one expired at 464 days, and the other did not progress at the end of study. Median is estimated using Kaplan-meier method. | 33 [33 to 33]

6. Other Pre Specified Outcome: Correlation of the Presence of PIK3CA Mutations in the Tumor With Time to Tumor Progression.
Description: Examining tumor tissue for PI3K mutations and correlating this statistically with clinical outcomes including time to tumor progression.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- 1PHIbA - Arm A - Cisplatin + GDC - 0941 Dose Level 1: Patients cohort 1 receive cisplatin and PI3K inhibitor GDC-0941. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients receive cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor: GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  If no patients in Cohort 1 experienced DLT's after 4 weeks, all patients in Cohort 2 will receive cisplatin and PI3K inhibitor GDC-0941, GDC-0941dose not to exceed 260mg.
  If 1 patient experiences a DLT in the first cohort, an additional cohort of 3 patients will be treated at the same dose level in cohort 2.
  If ≤1 patient has a DLT in 6 (cohort 1 and 2) treated at this same dose, this will be considered a tolerable dose to move to phase II.
- 2PHII 1 - Arm 1 - Cisplatin Only: Patients receive cisplatin in Arm I. Patients may crossover to Arm II upon disease progression.
  cisplatin:patients received cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients may crossover to Arm II upon disease progression.
  --------------------------------------------------------------------------------
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
- 2PHII2 - Arm 2 - Cisplatin and GDC-0941: Patients receive Cisplatin and PI3K inhibitor GDC-0941. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients received cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  patients receive PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  --------------------------------------------------------------------------------
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
  GDC -0941: Patients receive cisplatin as in Arm I and PI3K
- 2PHIICO - Crossover to Arm 2 - Cistplatin + GDC -0941: Crossover patient received Cisplatin and PI3K inhibitor GDC-0941 after found to have disease progression in Cisplatin only arm. Courses repeat in the absence of disease progression or unacceptable toxicity.
  cisplatin: patients received cisplatin IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  patient received PI3K inhibitor GDC-0941 orally (PO) one time a day (QD) on days 2-6, 9-13, 16-20, and 23-27. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  laboratory biomarker analysis: correlative studies
  pharmacological study: correlative studies
  dynamic contrast-enhanced MRI, diffusion-weighted MRI & chemical exchange saturation transfer MRI: correlative studies
Arm/Group | 1PHIbA - Arm A - Cisplatin + GDC - 0941 Dose Level 1 | 1PHIbB - Arm B - Cisplatin + GDC -0941 Dose Level -1 | 2PHII 1 - Arm 1 - Cisplatin Only | 2PHII2 - Arm 2 - Cisplatin and GDC-0941 | 2PHIICO - Crossover to Arm 2 - Cistplatin + GDC -0941
All-Cause Mortality (participants affected / at risk) | 6/6 | 0/0 | 1/2 | 2/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0 | 1/2 | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0 | 2/2 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1PHIbA - Arm A - Cisplatin + GDC - 0941 Dose Level 1 (N=6) | 1PHIbB - Arm B - Cisplatin + GDC -0941 Dose Level -1 (N=0) | 2PHII 1 - Arm 1 - Cisplatin Only (N=2) | 2PHII2 - Arm 2 - Cisplatin and GDC-0941 (N=3) | 2PHIICO - Crossover to Arm 2 - Cistplatin + GDC -0941 (N=1)
pericardial effusion (Cardiac disorders) | 0 | 0 | 0 (0) | 1 (1) | 0
paresthesia (Nervous system disorders) | 0 | 0 | 1 (1) | 0 (0) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1PHIbA - Arm A - Cisplatin + GDC - 0941 Dose Level 1 (N=6) | 1PHIbB - Arm B - Cisplatin + GDC -0941 Dose Level -1 (N=0) | 2PHII 1 - Arm 1 - Cisplatin Only (N=2) | 2PHII2 - Arm 2 - Cisplatin and GDC-0941 (N=3) | 2PHIICO - Crossover to Arm 2 - Cistplatin + GDC -0941 (N=1)
hypomagnesia (Metabolism and nutrition disorders) | 5 (10) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (3) | 3 (7) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gastroesophageal reflux disease (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
platelet count decreased (Investigations) | 3 (8) | 0 (0) | 1 (1) | 2 (5) | 0 (0)
white blood cell decreased (Investigations) | 3 (5) | 0 (0) | 0 (0) | 3 (13) | 0 (0)
neutrophil count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
acoustic nerve disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 1 (2) | 3 (6) | 1 (1)
fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (11) | 0 (0)
fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
hot flashes (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes